CLINICAL TRIAL: NCT04396457
Title: Phase 2 Study of Pembrolizumab Plus Pemetrexed for Elderly Patients With Non-squamous Non-small Cell Lung Cancer With PD-L1 Tumor Proportion Score of Less Than 50%: CJLSG1901
Brief Title: Pembrolizumab Plus Pemetrexed for Elderly Patients With Non-Sq NSCLC With PD-L1 < 50%: CJLSG1901
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Hospital Organization Nagoya Medical Center (Other)
Collaborators: Central Japan Lung Study Group (Unknown); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMC-CJLSG1901
Record Dates: First submitted 2020-01-14; First posted 2020-05-20 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Non-squamous Non-small-cell Lung Cancer; Cancer, Lung
MeSH Terms: conditions — Lung Neoplasms | interventions — pembrolizumab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab+Pemetrexed (Experimental): 200 mg of pembrolizumab is intravenously infused over 30 minutes and more on day 1.
  500 mg/m^2 of pemetrexed is intravenously infused over 10 minutes and more on day 1.
  *Administration of folic acid and vitamin B12 is started 1 week before the start of treatment with pemetrexed.
  And repeat the administration every 3 weeks as one cycle until the treatment cessation criteria are met. Upper limit of the pembrolizumab administration is 35 cycles, and the pemetrexed administration will continue until the treatment cessation criteria are met.
  Interventions: Drug: Pembrolizumab; Drug: Pemetrexed

INTERVENTIONS:
Drug: Pembrolizumab — Human PD-1 Monoclonal antibody
  Other Names: KEYTRUDA Injection
Drug: Pemetrexed — Antineoplastic antimetabolite
  Other Names: Alimta Injection

SUMMARY:
To evaluate the efficacy and safety of Pembrolizumab + Pemetrexed in elderly patients with non-squamous non-small cell lung cancer with Programmed cell death (PD) -ligand1 (L1) tumor proportion score (TPS) of less than 50%.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of Pembrolizumab + Pemetrexed in elderly patients with non-squamous non-small cell lung cancer with Programmed cell death (PD) -ligand1 (L1) tumor proportion score (TPS) of less than 50%.Primary endpoint is overall response rate and secondary endpoints are progression free survival (PFS), 1 year PFS rate, overall survival and adverse event.

ELIGIBILITY:
Inclusion Criteria:

1. Non-squamous non-small cell lung cancer (NSCLC) confirmed by histology or cytology.
2. Not received prior systemic treatment with stage IV, or recurrent NSCLC. Subjects who received adjuvant therapy are eligible if the adjuvant therapy was completed at least 12 months prior to the development of metastatic disease.
3. PD-L1 TPS of less than 50% with 22C3 antibody.
4. With at least one measurable lesion based on RECIST 1.1.
5. Age of 75 years or older on the day of informed consent.
6. ECOG Performance Status 0-1.
7. Without activating mutation in EGFR or ALK chromosomal translocation.
8. Absence of severe impairments of major organs.
9. Life expectancy of 12 weeks or more from the treatment start date.
10. Prior to the study registration, able to provide written informed consent after a thorough explanation of the study content.

Exclusion Criteria:

1. Before the first dose of trial treatment:

   Had major surgery (<3 weeks prior to the first dose)
2. Received radiation therapy to the lung that exceeds 30 Gy within 6 months of the first dose of the study treatment.
3. Completed palliative radiotherapy within 7 days of the first dose of the treatment.
4. Has received a live-virus vaccination within 30 days of planned treatment initiation.

   Seasonal flu vaccines that do not contain live virus are permitted.
5. Has clinically active diverticulitis, intra-abdominal abscess, GI obstruction, peritoneal carcinomatosis.
6. Has a history of malignancy except if the subject has undergone curative therapy without recurrence for 5 years since initiation of that therapy.
7. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
8. Previously had a severe hypersensitivity reaction to treatment with another mAb.
9. Has a known sensitivity to any component of pemetrexed
10. Has active autoimmune disease that has required systemic treatment in past 2 years
11. Is on chronic systemic steroids. Subjects with asthma that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections would not be excluded from the study.
12. Is unable to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs), other than an aspirin.
13. Is unable or unwilling to take folic acid or vitamin B12 supplementation.
14. Had prior treatment with any other anti-PD-1, or PD-L1 or PD-L2 agent or an antibody targeting other immuno-regulatory receptors or mechanisms.
15. Has an active infection requiring therapy.
16. Has a history of Human Immunodeficiency Virus (HIV)
17. Has known active Hepatitis B or C. Active Hepatitis B is defined as a known positive HBsAg result.
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the Principal Investigator.
19. Has symptomatic ascites or pleural effusion.
20. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
21. Patients wishing their partner to become pregnant during the study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-05-25 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to approximately 3 years
  Overall response rate

SECONDARY OUTCOMES:
Progression free survival | Up to approximately 3 years
  Progression free survival
1 year progression free survival rate | 1 year
  1 year progression free survival rate
Overall survival | Up to approximately 3 years
  Overall survival
Adverse event | Up to approximately 3 years
  Adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihito Kogure, MD, PhD, Principal Investigator — National Hospital Organization Nagoya Medical Center
Locations (1):
- National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kogure Y, Hashimoto H, Daga H, Fukuda Y, Bessho A, Yamada T, Toi Y, Kimura T, Yoshioka H, Azuma K, Furuya N, Fukui Y, Saito AM, Yamamoto N, Saka H, Kondo M. Pembrolizumab and Pemetrexed for Older Patients With Nonsquamous NSCLC and Programmed Cell Death-Ligand 1 Tumor Proportion Scores of Less Than 50. JTO Clin Res Rep. 2024 Dec 24;6(3):100784. doi: 10.1016/j.jtocrr.2024.100784. eCollection 2025 Mar. PMID 40007549